CLINICAL TRIAL: NCT01676428
Title: A Pilot Study of Focal Ablative STereotactic RAdiosurgery for Cancers of the Kidney or Isolated Adrenal Metastases
Acronym: FASTRACK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peter MacCallum Cancer Centre, Australia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11/106; U1111-1132-5574 (Registry Identifier: ANZCTR)
Record Dates: First submitted 2012-08-14; First posted 2012-08-31 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-03

CONDITIONS: Cancer
Keywords: Kidney; Renal; Radiotherapy; Stereotactic; Cancer
MeSH Terms: conditions — Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Radiotherapy (Experimental): The interventional treatment will be prescribed as a 2-tiered dose scheduled dependant of target size.
  For lesions <5cm, a single fraction of 26 Gy will be prescribed. For lesions ≥5cm a fractionated course of 15Gy by 3 fractions will be prescribed, delivered at least 48 hours apart.
  Interventions: Radiation: Radiotherapy

INTERVENTIONS:
Radiation: Radiotherapy — The investigational treatment will be prescribed as a 2-tiered dose scheduled dependant on target size.
  For lesions <5cm, a single fraction of 26Gy will be prescribed. For lesions ≥5cm a fractionated course of 14Gy by 3 fractions will be prescribed, delivered at least 48 hours apart.

SUMMARY:
This is a "proof of concept" study, to assess the feasibility of introducing a novel high-precision radiotherapy technique called "stereotactic radiosurgery" (SRS) or "stereotactic body radiotherapy" (SBRT) for the treatment of kidney cancers in Australia. This study aims to invite 20 patients with renal cell carcinoma and 10 patients with isolated adrenal metastases from non-small cell carcinoma who are either medically inoperable, high risk for surgery, or decline surgery to participate. In cohort of patients with renal cell carcinoma, both patients with primary disease only, and those patients who have limited metastases (≤5) will be eligible. Besides technical feasibility of delivering this treatment, this study will be to assess efficacy, toxicity and tumour response using a novel imaging biomarker called diffusion weighted-MRI.

DETAILED DESCRIPTION:
FASTRACK is a 2 -cohort, non-randomised prospective feasibility study. Anticipated total duration of accrual is approximately 24 months, with all patients expected to complete all protocol treatment and imaging within a further 3 months. The trial will close after the last patient has completed his/her last protocol related follow-up visit (at 12 months post-treatment).

Cohort 1: patients with renal cell carcinoma within the kidney Cohort 2: patients with solitary adrenal metastases from non-small cell lung carcinoma The investigational treatment will be prescribed the covering isodose, ensuring that 99% of the PTV is covered by 100% of the dose (D99=100%). It is anticipated that most treatments should be highly conformal. Treatment must be delivered with at least six (6) non-opposing conformal megavoltage photon beams. It is anticipated that a typical range of beam numbers would be 8 to 12, comprising of at least 6 co-planar beams and 1-2 non-coplanar beams. No cytotoxic chemotherapy is allowed within 3 weeks or concurrently with respect to the investigational treatment. Consultation with the treating radiation oncologist is strongly recommended if chemotherapy is to be considered after the investigational treatment and before documented disease progression, to prevent unforeseen combined toxicities. Targeted agents (such as sunitinib) are exempt from this recommendation.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* All patients must have radiological diagnosis or biopsy confirmed diagnosis of either:

  1. Cohort 1: renal cell carcinoma with a single lesion within kidney, or with primary kidney tumour intact and no more than 5 documented metastases, or
  2. Cohort 2: single adrenal metastases with extra-adrenal disease controlled
* ECOG performance of 0-2 inclusive.
* Either medically inoperable, technically high risk for surgery or decline surgery.
* Informed consent.

Exclusion Criteria:

* Cytotoxic chemotherapy within 3 weeks of commencement of treatment, or concurrently with treatment. Delivery of targeted agents (such as sunitinib) are allowable only when at least 7 days separate the delivery of the proposed agent and the delivery of the stereotactic radiotherapy.
* Previous high-dose radiotherapy to upper abdomen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2012-05; Primary Completion 2014-10 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
The number of patients who complete prescribed treatment. | After 24 months
  This is defined as patients who successfully receive the treatment plan as prescribed, achieving all nominated dose constraints, and are able to tolerate the treatment(s)

SECONDARY OUTCOMES:
Toxicity of SBRT in study patients measured using CTCAE V4.0 | Between 2-4 weeks after radiotherapy and 3 monthly for 12 months
  Specific toxicities will include, but are not limited to;
  * Gastrointestinal (Nausea, vomiting, diarrhoea, acute ulceration)
  * Pulmonary (atelectasis, cough, dyspnoea, hypoxia, pleural effusion, fibrosis)
  * Skin/chest wall (radiation dermatitis, rib fracture)
  * Kidney (acute renal dysfunction) Freedom from severe toxicity will be reported asn defined as: time from treatment delivery until first recorded grade 4, or 5 toxicity as measured by CTCAE V4.0.
Efficacy of stereotactic radiosurgery | 1 year after treatment
  Effective SBRT is defined as a treatment which results in local control at 1 year after treatment. Local control is defined as lack of progression of the target lesion as measured by RECIST criteria. RECIST criteria are a CT evaluation of change in tumour size.
Feasibility of using Diffusion weighted-MRI for response assessment. | At Baseline, 14 days (+/-3 days) and at the definitive response assessment (70days +/-10days)
  Feasibility will be measured by the quality of image of the diffusion weighted-MRI recorded by the investigating radiologists.

CONTACTS AND LOCATIONS:
Overall Officials: Shankar Siva, Principal Investigator — Peter MacCallum Cancer Centre, Australia
Locations (1):
- Peter MacCallum Cancer Centre, East Melbourne, Victoria, Australia

REFERENCES:
- [Derived] Pham D, Thompson A, Kron T, Foroudi F, Kolsky MS, Devereux T, Lim A, Siva S. Stereotactic ablative body radiation therapy for primary kidney cancer: a 3-dimensional conformal technique associated with low rates of early toxicity. Int J Radiat Oncol Biol Phys. 2014 Dec 1;90(5):1061-8. doi: 10.1016/j.ijrobp.2014.07.043. Epub 2014 Oct 13. PMID 25442039